CLINICAL TRIAL: NCT04891718
Title: A Phase 0 Master Protocol Using the CIVO® Platform to Evaluate Intratumoural Microdoses of Anti-Cancer Therapies in Patients With Solid Tumours
Brief Title: CIVO Intratumoural Microdosing of Anti-Cancer Therapies in Australia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Termination by pharmaceutical sponsor
Sponsor: Presage Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBI-MST-02
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumour
Keywords: HNSCC; SCCHN; lymphoma; sarcoma; breast adenocarcinoma; melanoma; intratumoural microdosing; microdose injection; microdosing; in vivo oncology; in vivo drug sensitivity; tumour microenvironment; multiplexed immunohistochemistry; head and neck cancer; pharmacodynamic biomarkers; CIVO; master protocol; precision oncology
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoma; Sarcoma; Melanoma; Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This Master Protocol is designed as an umbrella concept trial for the ongoing evaluation of multiple agents in individual CIVO Phase 0 substudies. Each substudy is considered an "Experimental Arm" with specified investigational agents and combinations to be evaluated. Comparisons will not be made between experimental arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MVC-101 and Nivolumab (Experimental): Patients with HNSCC who are scheduled for surgical biopsy or tumour resection surgery will be injected at least four hours to up to three days prior to surgery using the CIVO device. Each needle of the CIVO device will deliver up to 8.3 microliters of solution, including a vehicle control (sterile saline and solution stabilizer), a pre-cleaved/pre-activated drug control (cMVC-101), MVC-101 (the prodrug), or nivolumab as single agents or as combinations. Each drug will be delivered in subtherapeutic microdoses, and each microdose is simultaneously injected in a columnar fashion through each of 3, 5, or 8 needles (in a device configuration determined by tumour dimensions) into a single solid tumour or effaced metastatic lymph node.
  Interventions: Biological: MVC-101; Biological: Nivolumab; Combination Product: MVC-101 + Nivolumab

INTERVENTIONS:
Biological: MVC-101 — Intratumoural microdose injection by the CIVO device.
  Other Names: TAK-186
Biological: Nivolumab — Intratumoural microdose injection by the CIVO device.
  Other Names: Opdivo; BMS-936558
Combination Product: MVC-101 + Nivolumab — Intratumoural microdose injection by the CIVO device.

SUMMARY:
This is a multi-center, open-label Phase 0 Master Protocol in Australia designed to study the localized pharmacodynamics (PD) of anti-cancer therapies within the tumour microenvironment (TME) when administered intratumourally in microdose quantities via the CIVO device in patients with surface accessible solid tumours for which there is a scheduled surgical intervention. CIVO stands for Comparative In Vivo Oncology. Multiple substudies will include specified investigational agents and combinations to be evaluated.

DETAILED DESCRIPTION:
CIVO is a research tool composed of a hand-held single-use sterile injector coupled with fluorescent tracking microspheres called CIVO GLO that mark the sites of drug microdose injection, enabling rapid assessment of multiple oncology drugs or drug combinations simultaneously within a patient's tumour. Tumour responses to cancer treatments are highly context-specific and often involve complex interactions between the anti-cancer therapy, genetically diverse tumour cells, and a heterogeneous TME. This complexity is rarely modeled accurately in preclinical translational models of cancer. By utilizing intratumoural microdose injections with CIVO in advance of scheduled surgical intervention, this study will evaluate anti-cancer therapies directly in patients each with their own unique tumour genomic profile, intact TME, and immune system functional status. Because the platform delivers microdose amounts of each test agent or combination directly into the patient's tumour tissue, hypotheses can be tested earlier in the drug development process.

The CIVO device penetrates solid tumours and simultaneously delivers subtherapeutic microdoses of up to eight anti-cancer agents or combinations of anti-cancer agents co-injected with CIVO GLO into discrete regions of the tumour as drug columns. At the time of the planned surgical intervention (at least four hours to up to seven days after the CIVO microdose injection), the injected tumour tissue is then excised and tumour responses are assessed via histological staining of tumour cross-sections sampled perpendicular to each injection column. Co-injection with CIVO GLO enables identification of each injection site during resection as well as in tissues stained for analysis. This Phase 0 Master Protocol is aimed at distinguishing promising candidates earlier in the drug development process while also avoiding systemic toxicities associated with typical clinical exposures to these therapies.

ELIGIBILITY:
*This list is representative of study inclusion/exclusion criteria. Each substudy may include variations on these criteria.

Inclusion Criteria:

1. Ability and willingness to comply with the study's visit and assessment schedule.
2. Male or female ≥ 18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of [solid tumours] indicated in the relevant substudy(ies).
4. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. At least one lesion (primary tumour, recurrent tumour, or effaced metastatic lymph node) ≥ 2 cm in the shortest diameter that is surface accessible for CIVO injection that may be guided by ultrasound if appropriate and for which there is a planned surgical intervention. Treatment plan may include adjuvant radiation or chemotherapy and patients should have no medical contraindication to surgery.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * Are of childbearing potential who agree to practice a highly effective method of contraception from the time of signing the Informed Consent Form (ICF) and during study participation OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from donating ova during study participation.

Male patients, even if surgically sterile (i.e., status post-vasectomy), who:

* Agree to practice effective barrier contraception from the time of signing the ICF and during study participation OR agree to completely abstain from heterosexual intercourse.
* Agree to refrain from donating sperm during study participation.

Exclusion Criteria:

1. Tumours or effaced nodes that are anticipated by the Investigator to lack a sufficient volume of viable tumour tissue (based on available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports) for CIVO injection due to size, location, necrosis, cysts, excessive stroma, fibrosis, or treatment-induced tissue changes.
2. Tumours near or involving critical structures for which, in the opinion of the treating clinician, injection would pose undue risk to the patient.
3. Female patients who are:

   * Breastfeeding
   * Have a positive β-subunit human chorionic gonadotropin (β-hCG) pregnancy test at screening verified by the Investigator.
4. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.
5. Patients with a history of concurrent second cancers requiring active, ongoing systemic treatment.
6. Patients with active autoimmune diseases requiring treatment.
7. Patients that have received a live vaccine within 4 weeks of the baseline/screening visit.
8. Use of any of the following ≤ 2 weeks prior to CIVO injection:

   1. Chronic systemic immunosuppressive therapy or corticosteroids (e.g., prednisone or equivalent exceeding a total dose of 140 mg over the last 14 days). Intranasal, inhaled, topical, or local corticosteroid injections (e.g., intra-articular injection), or steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) are exceptions to this criterion.
   2. Biological response modifiers for treatment of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Quantification of Cell Death and Immune Cell Biomarkers by IHC and In-Situ Hybridization | 4 hours-7 days after microdose injection
  Quantification of biomarker-positive and biomarker-negative cells will be performed within the tumour microenvironment around each of the injection sites in each resected patient sample by IHC and ISH. An aggregate analysis of this quantification may be done across patient samples in each substudy to evaluate trends in tumour response. The biomarkers evaluated may include, but are not limited to biomarkers for cell death (e.g. cleaved caspase 3), T-cells (e.g. CD3, CD8/Granzyme B, CD4), natural killer (NK)/myeloid cells (e.g. CD56/Granzyme B, CD86, CD68, CD163), and proinflammatory cytokines (e.g., interferon gamma, tumour necrosis factor alpha, interferon gamma-induced protein 10).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | Up to 28 days after microdose injection
  Relationship of AE to study drug(s) or CIVO device will be determined using an AE Relatedness Grading System.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Presage Biosciences
Locations (3):
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571